CLINICAL TRIAL: NCT06399562
Title: Related Factors of Hp Infection in Physical Examination and Community Population in Hunan Province: A Cross-sectional Study
Brief Title: Related Factors of Hp Infection in Physical Examination and Community Population in Hunan Province
Status: Completed | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: The Second People's Hospital of Huaihua (Unknown); Yueyang Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Fen Wang, Professor, The Third Xiangya Hospital of Central South University
Other Study IDs: FastI 22136
Record Dates: First submitted 2024-04-20; First posted 2024-05-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the physical examination population: the physical examination population from the health management center of the Third Xiangya Hospital
  Interventions: Diagnostic Test: carbon-13 urea breath test (13C-UBT); Behavioral: questionnaires
- the community residents: the family-based community residents in Changsha
  Interventions: Diagnostic Test: carbon-13 urea breath test (13C-UBT); Behavioral: questionnaires

INTERVENTIONS:
Diagnostic Test: carbon-13 urea breath test (13C-UBT) — The H. pylori infection was detected by carbon-13 urea breath test (13C-UBT), a delta over baseline (DOB) of ≥4.0 was considered positive for H. pylori, and a DOB<4.0 was considered negative.
Behavioral: questionnaires — The related factors of H. pylori infection were investigated by questionnaire survey. The physical examination population participated in the questionnaires of the physical examination center, which included basic demographic characteristics and living habits, and filled out the questionnaires on the use of serving chopsticks at the same time. In the community, members of each eligible family were asked to complete a questionnaire including the details such family general information, basic information of every family member, personal living habits, past medical history, and so on.

SUMMARY:
This study intends to investigate the prevalence and risk factors of Helicobacter pylori (H. pylori) infection in the population of physical examination centers and communities. The physical examination population from the health management center of the Third Xiangya Hospital and the family-based community residents in Changsha were randomly selected. The H. pylori infection was detected by carbon-13 urea breath test (13C-UBT), and the related factors of H. pylori infection were investigated by questionnaire survey. The study provides supporting evidences to implement family-base H. pylori management to curb its intrafamilial spread. The results have important clinical implications in refinement of eradication strategies and impact on public health policy formulation for related disease prevention.

ELIGIBILITY:
Inclusion Criteria:

1. population aged 4-90 years, no requirement for gender;
2. the physical examination population from the health management center of the Third Xiangya Hospital;
3. the family-based community residents in Changsha City [families containing two or more family members (living together for more than 10 consecutive months per year) and the family members aged 3 years and above];

Exclusion Criteria:

1. people with use of antibiotics, bismuth or Chinese traditional medicines with antibacterial effects in the previous 4 weeks of 13C-UBT, or H2 receptor antagonists, PPIs, P-CAB or other drugs affecting H. pylori activity within the previous 2 weeks of 13C-UBT;
2. people with H. pylori treatment within the past 3 months;
3. People who fasted less than 3 hours before 13C-UBT;
4. people with other contraindications to performing 13C-UBT;
5. people living alone in a family;
6. people with incomplete questionnaire information;
7. people with serious diseases or clinical conditions that may interfere with the evaluation of the results of the study, such as severe heart, liver, lung, and renal insufficiency, low immunity, and so on;
8. people with mental illness and communication disorders;
9. people deemed unsuitable by the researchers to participate in this project;

Ages: 4 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 1. the physical examination population from all over the country was randomly selected from the Health Management Center of the Third Xiangya Hospital;
  2. the family-based community residents were randomly selected in Changsha. [families containing two or more family members (living together for more than 10 consecutive months per year) and the family members aged 3 years and above];
Sampling Method: Non-Probability Sample
Enrollment: 1516 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | through study completion, an average of 1 week
  carbon-13 urea breath test

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient department of gastroenterology of the Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No